CLINICAL TRIAL: NCT07224503
Title: Phase II Randomized Controlled Trial of C-SMART Versus BE Well for Patients With Brain Tumors on Neurocognitive and Neuroimaging Outcomes
Brief Title: C-SMART vs BE Well for Patients With Brain Tumors
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Labs for intervention not currently open
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Psychological Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MCC-25-22557; HM300000218 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Strategies, Mindfulness, and Rehabilitation Therapy (C-SMART) (Experimental): Modular tele-neuropsychological rehabilitation blending both cognitive rehabilitation with integrated mindfulness meditation training.
  Interventions: Behavioral: C-SMART
- Brain health Education and Wellness (BE Well) (Active Comparator): Time-matched educational videos focused on maximizing brain health in the context of brain tumor.
  Interventions: Behavioral: BE Well

INTERVENTIONS:
Behavioral: C-SMART — Eight weekly, 45-60 minute, 1:1 tele-intervention sessions, targeting neurocognitive weaknesses identified from baseline cognitive testing
  Arms: Cognitive Strategies, Mindfulness, and Rehabilitation Therapy (C-SMART)
Behavioral: BE Well — Eight weekly 45- to 60-minute video lectures
  Arms: Brain health Education and Wellness (BE Well)

SUMMARY:
The goal of this clinical trial is to learn about the acceptability and feasibility of Cognitive Strategies, Mindfulness, and Rehabilitation Therapy (C-SMART) and Brain health Education and Wellness (BE Well) in adults with brain tumors and their caregivers.

Participants will be assigned to one of the two groups:

* Cognitive Strategies, Mindfulness, and Rehabilitation Therapy (C-SMART) is a recently developed virtual intervention combining both cognitive rehabilitation with mindfulness meditation training. The manualized program consists of 8 weekly 1:1 tele intervention sessions, targeting cognitive weaknesses identified from baseline cognitive testing.
* Brain health Education and Wellness (BE Well) intervention consists of 8 weekly videos focused on maximizing brain health in the context of brain tumor.

Participants will also be asked to:

* participate in two in-person visits involving an MRI and neurocognitive tests
* complete a survey the the beginning and end of the study
* if in BE Well group, answer a few questions after watching each video

ELIGIBILITY:
Patient Inclusion Criteria:

* Patient of Virginia Commonwealth University Neuro-Oncology clinic
* Confirmed primary brain tumor diagnosis by histology or neuro-oncologist review of imaging
* At least one domain of neurocognitive function >1.5 SD below the average or the individual's estimated premorbid functioning, using the expanded International Cognition and Cancer Task Force (ICCTF) clinical trials battery and Test of Premorbid Functioning62 for comparison; (3) >1 month post brain surgery and/or radiation therapy, if applicable;
* Estimated premorbid intelligence >75.
* Patients must be age 18+ and
* Primarily English speaking.

Patient Exclusion Criteria:

* Presence of major neurocognitive impairment that would prevent participation in the intervention, and/or severe aphasia, and/or inability to understand and provide informed consent
* Inability to attend weekly telehealth appointments
* Clinically significant insomnia symptoms coupled with report that insomnia is more interfering than cognitive symptoms
* < 1 month post brain surgery and/or radiation therapy
* Unstable internet connection or an inability to work teleconferencing software. Participants will be supplied an iPad if they do not have an adequate device.
* Participants cannot have metal in their body as the MRI scan could cause them harm
* If female of childbearing years, they cannot be pregnant as the MRI scan may pose risk to the unborn fetus

Caregiver Inclusion Criteria

* Must enroll with a patient (see criteria above)
* Must be age 18+ and
* Primarily English speaking

Caregiver Exclusion Criteria

-N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Assess the feasibility of the C-SMART and BE Well protocols in brain tumor patients and caregivers- Eligibility Rate | From time participant indicates interest to screening completion, 4 weeks
  The percentage of participants that are eligible to enroll
Assess the feasibility of the C-SMART and BE Well protocols in brain tumor patients and caregivers- Enrollment Rate | From screening to intervention initiation, 8 weeks
  The percentage of participants that enroll
Assess the feasibility of the C-SMART and BE Well protocols in brain tumor patients and caregivers -- retention rate | From baseline to end of study, 28 weeks
  The percentage of participants that complete the post-intervention data collection
Assess the acceptability of the C-SMART and BE Well protocols in brain tumor patients and caregivers -- intervention completion rate | From baseline to end of intervention, 16 weeks
  The percentage of participants that complete the the protocol assigned interventions
Assess the acceptability of the C-SMART and BE Well protocols in brain tumor patients and caregivers- Participant satisfaction ratings | From baseline to post-intervention survey completion, 20 weeks
  Participant ratings of satisfaction. Participants will rate the following questions on a scale from completely disagree to completely agree: C-SMART/BE Well Meets my approval; C-SMART/BE Well is appealing to the patient; "I like C-SMART/BE Well"; "I welcome C-SMART/BE Well". Additionally, participants will answer the following question on a scale from extremely dissatisfied to extremely satisfied: "When you signed up for the study, you were told that you would be randomized to either C-SMART or BE Well Videos. How satisfied are you with the group you were randomized to?"
Assess the acceptability of the C-SMART and BE Well protocols in brain tumor patients and caregivers- Participant recommendation ratings. | From baseline to post-intervention survey completion, 20 weeks
  Participant ratings of intervention recommendation Participants will answer the following question: Would "you" (the patient) recommend C-SMART/BE Well to other brain tumor patients?

SECONDARY OUTCOMES:
Investigate effect of interventions on neurocognitive tests Hopkins Verbal Learning Test (verbal learning and memory) | Baseline to post-intervention assessment, up to 28 weeks
  Changes in neurocognitive assessment scores (pre vs post intervention) between groups based on the Hopkins Verbal Learning Test (verbal learning and memory) neurocognitive test. Participant performance on the verbal learning and memory task will consist of three learning trials and a delay. A high score on the learning trials but a very low score on the delayed recall would show that the person can learn but has difficulty retrieving previously learned information.
Investigate effect of interventions on neurocognitive test Controlled Oral Word Association (verbal fluency) | Baseline to post-intervention assessment, up to 28 weeks
  Changes in neurocognitive assessment scores (pre vs post intervention) between groups based on the Controlled Oral Word Association (verbal fluency) neurocognitive test. Participant performance on the verbal fluency task will consist of generating words in 60 seconds on phonemic trials (words that start with a specific letter) and semantic trials (words that fall into a specific category). Scores are the number of correctly retrieved words. A higher raw score indicates greater verbal fluency.
Investigate effect of interventions on neurocognitive test Trail Making (attention and task switching) | Baseline to post-intervention assessment, up to 28 weeks
  Changes in neurocognitive assessment scores (pre vs post intervention) between groups based on Trail Making (processing speed and task switching). Participant performance will consist of time (in seconds) to complete a processing speed and switching task in which participants are asked to draw lines in sequential order, and then switch between two overlearned sequences. A shorter time to completion would indicate greater processing speed and task switching.
Investigate effect of interventions on neurocognitive test | Baseline to post-intervention assessment, up to 28 weeks
  Changes in neurocognitive assessment scores (pre vs post intervention) between groups based on the Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV) Processing Speed Index (processing speed). Participant performance on the processing task will consist of indicating matching symbols and drawing symbols linked to numbers based on a key. The score is the number of completed items during 120 seconds. A higher raw score indicates faster processing speed.
Investigate effect of interventions on neurocognitive test WAIS-IV Digit Span Tests (auditory working memory) | Baseline to post-intervention assessment, up to 28 weeks
  Changes in neurocognitive assessment scores (pre vs post intervention) between groups based on the Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV) Digit Span Tests (auditory working memory). Participant performance on the working memory task will consist of repeating back a string of numbers in order, in reverse order, and then in ascending order -- after every two trials completed correctly, the number increases by one-digit. Scores are the number of items completed correctly. A higher raw score indicates greater working memory.
Investigate effect of interventions on neurocognitive test Neuropsychological Assessment Battery Naming Test (naming abilities) | Baseline to post-intervention assessment, up to 28 weeks
  Changes in neurocognitive assessment scores (pre vs post intervention) between groups based on the Neuropsychological Assessment Battery Naming Test (naming abilities). Participant performance on the naming task will consist of naming pictured objects. A higher raw score indicates greater expressive language and naming abilities.
Investigate effect of interventions on neurocognitive test Delis-Kaplan Executive Function System Color-Word Inference Test (inhibition and switching) | Baseline to post-intervention assessment, up to 28 weeks
  Changes in neurocognitive assessment scores (pre vs post intervention) between groups based on the Delis-Kaplan Executive Function System Color-Word Inference Test (inhibition and switching). Participant performance on the inhibition and switching task consists of reading words and naming the color of words in order and while switching between the two. Scores are the time it takes to complete each trial.
Investigate effect of interventions on subjective cognition | Baseline to post-intervention assessment, up to 20 weeks
  Changes in subjective cognition (pre vs post intervention) between groups based on the Neuro-Qol Short Form the National Institutes of Health (NIH) toolbox. Participants rate their experience of cognitive slips on 4 questions from "never" to "very often", and 4 questions from "no difficulty" to "cannot do". Higher scores indicate greater subjective cognition. Scores range from 8-40. Raw scores can be converted into standardized scores (T-scores) with a mean of 50 and a standard deviation (SD) of 10. Thus, a person who has a T-score of 60 is one SD above the average of the US general population.
Investigate effect of interventions on fatigue | Baseline to post-intervention assessment, up to 20 weeks
  Changes in fatigue (pre vs post intervention) between groups based on the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue short form. Participants rate their experience of fatigue on 4 items from "not at all" to "very much". Higher scores indicate greater fatigue. Scores range from 4-20. Raw scores can be converted into standardized scores (T-scores) with a mean of 50 and a standard deviation (SD) of 10. Thus, a person who has a T-score of 60 is one SD above the average of the US general population.
Structural brain changes | From baseline to post-outcome assessment, 28 weeks
  Change in brain volume (pre vs. post intervention) between groups based on brain imaging (MRI) data. The volume of lateral ventricle in the hemisphere opposite to the tumor will be measured, using 3D Slicer (https://www.slicer.org) to calculate the ventricular volume at each time point which will serve as an index of diffuse cerebral volume loss.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Braun, Ph.D, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual patient data "IPD" at this time.